CLINICAL TRIAL: NCT03700060
Title: Communication and Compliance With Guidelines for Antibiotic Prescribing by General Practice to Nursing Home Residents With Suspected Urinary Tract Infections -A Research Protocol for a Cross-Sectional Study in the Primary Care Sector
Brief Title: Communication and Compliance for Antibiotic Prescribing by General Practice to Nursing Home Residents With Suspected UTI
Status: Completed | Type: Observational
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Responsible Party: Principal Investigator, Sif Helene Arnold, Principal Investigator, Research Unit Of General Practice, Copenhagen
Other Study IDs: UTI in nursing homes
Record Dates: First submitted 2018-04-09; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Urinary Tract Infections; Communication; Compliance, Medication
MeSH Terms: conditions — Urinary Tract Infections; Communication; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Practice: Volunteering General Practices who registers contacts from nursing homes on residents with suspected UTI

SUMMARY:
Antibiotic resistance is becoming a bigger problem. If the problem remains unsolved, the WHO predicts a return to the pre-antibiotic era. Overtreatment with antibiotics drives development of resistant bacteria and adverse events in patients, thus identification and rectifying factors leading to unnecessary antibiotic prescriptions are a public health problem.

Urinary Tract Infections (UTIs) are the most commonly diagnosed infection in nursing homes (NH). A prevalence study showed that in up to 76% of all antibiotic prescriptions in Danish NHs the indication was UTI. In this particular group of patients with suspected UTI, the literature has repeatedly shown that a vast amount of these antibiotic courses are inappropriate.

As people age, the prevalence of asymptomatic bacteriuria increases significantly. Asymptomatic bacteriuria is a condition that should not be treated with antibiotics. Thus, the treatment decision in this group should not rely on the result of urinary testing and should only commence, when classical urinary symptoms are present. Urinary testing of NH residents is one of the drivers of overtreatment. Therefore, a recent Danish guideline from Institute of Rational Pharmacology (IRF) on elderly with suspected UTI suggest that urine culture should only be performed when typical urinary symptoms are present and that antibiotic prescribing should be delayed until the result of the culture is available whenever possible. It is unknown to what extent Danish GPs follows these guidelines.

NH residents are often immobile, therefore; the diagnostic process of UTI in NH residents differs from the norm, which could also explain some part of the inappropriate prescribing. Immobility introduces physical distance between patient and GP because the patient is unable to visit the General Practitioners office. Because home visits are rare, when a UTI is suspected, NH staff usually contacts the GP in writing, over the phone and occasionally in person to relate the patient history and physical findings.

When another link in the communication chain between patient and GP is added, clinical information passes through additional health professionals and the risk of communication error and misunderstanding increases. Some forms of communications may be more suited to fit this setting than others. When communicating in person, it is possible to take non-verbal cues into account and immediately clear up insecurities. Communication by phone eliminates non-verbal cues, but a dialog about unclarified aspects is still attainable. Written communication, however, has none of the clarifying traits of the former, and to elaborate on the content the GP will have to contact the NH, which takes time in an already packed schedule.

The investigators hypothesize that the more direct the contact form, the better the quality of clinical information, which leads to increased compliance with guidelines. Thus by proxy, our hypothesis becomes that compliance to guidelines increases with directness of contact form. The aim of this study is to investigate to which degree the guidelines on antibiotic prescribing for NH residents with suspected UTI are followed and how the communication form affects adherence to guidelines.

ELIGIBILITY:
Inclusion Criteria:

* The general practices included in this study must all be from the Capital Region of Denmark.
* Each practice must have as many patients in the target population that an estimated five registered contacts during the registration period is feasible.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nursing Home residents, who are living permanently in a nursing home and exhibits signs or symptoms of acute UTI according to themselves, nursing home staff or the GP
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
How many suspected UTIs in nursing home residents are treated in accordance with guidelines? | 3rd of april - 30th of june
  For each suspected UTI, it must be determined if the GP handles the patient according to guidelines. The answer to this question will be in percent of all suspected UTIs with a subanalysis of why the reason why they are not treated in accordance (e.g. no urinary symptoms)

SECONDARY OUTCOMES:
Is mode of communication associated compliance to the guideline? | 3rd of april - 30th of june
  A logistic regression model will be developed, where the outcome variable states if the suspected UTI is treated according to the guideline or not. The dependent variables are contact form from nursing home to GP and contact form from GP to nursing home.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit of General Practice, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The IPD is anonomous when it leaves the General Practice and can therefore freely be shared with other researchers. The project group will register the protocol on clinicaltrial.gov and publish research papers on the collected data.